CLINICAL TRIAL: NCT05382000
Title: Evaluation of an Advanced Triage Tool for Gynecology and Obstetrics Emergencies Based on Artificial Intelligence Algorithms
Brief Title: Artificial Intelligence (IA) Advanced Triage Tool for G&O Emergencies
Acronym: TIAGO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-TIA-2021-81
Record Dates: First submitted 2022-04-28; First posted 2022-05-19 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Once the patient's consent has been obtained, the patient will be assessed sequentially in the same triage space. Initially, a nurse will classify the patient in the triage box using the MAT system according to the usual practice. Then, another professional from the center, trained in the use of the Mediktor Hospital ® tool, and who has not been present in the conventional sorting, will perform the advanced IA triage in the same space, both professionals being blind to the result of each of the tools.
  Attention in the Emergency Service Once the sequential triage is completed, the patient will return to the Gynecology and Obstetrics Emergency Room. The patient's care will be performed according to usual clinical practice, following the triage assessment performed with the MAT system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Inclusion in the study will be proposed to all patients who come to the Emergency Department of the Gynecology and Obstetrics Service
  The planned procedures for this group are as follows:
  1. Obtaining informed consent.
  2. Sequential triage - Patients will be evaluated sequentially using the MAT system according to standard practice. Next, another professional from the center, trained in the use of the Mediktor Hospital ® tool, will perform the advanced triage in the same space, both professionals being blind to the result of each of the tools.
  3. Once the sequential triage is finished, the patient's care will be carried out according to usual clinical practice, following the triage assessment carried out with the MAT system.
  4. Retrieval and introduction of data in DRF - Data of the study variables will be retrieved from the emergency report issued in the Gynecology and Obstetrics Emergency area and will be entered into an electronic DRF for subsequent analysis and processing.
  Interventions: Diagnostic Test: Advanced triage tool for Gynecology and Obstetrics emergencies based on artificial intelligence algorithms.

INTERVENTIONS:
Diagnostic Test: Advanced triage tool for Gynecology and Obstetrics emergencies based on artificial intelligence algorithms. — After the conventional triage, a second independent doctor will make the suit with the Mediktor Hospital tool.. In less than 3 minutes and with an average of 14 questions, Mediktor performs an interrogation very similar to what an emergency doctor would do. The professional version allows the health professional to modify the course of the questions in the middle of the evaluation, if he considers it necessary to go deeper into some aspect of the anamnesis. The system allows you to see in real time the diseases that Mediktor considers possible during the evaluation.
  At the end of the triage process, Mediktor offers the level of urgency and a list of possible diagnoses based on the signs and symptoms answered. The professional can change the level of urgency if he considers it beneficial for the patient.
  Once the two triages (Conventional and Mediktor) have been carried out, the patient will be seen according to the care protocols of the center.

SUMMARY:
Triage represents the first opportunity to classify patients who come to an Emergency Department (ED) and to be able to identify, prioritize high-risk patients and efficiently allocate the limited resources that are available. Therefore, the purpose of triage in the ED is to prioritize patients, detecting those that are urgent (that cannot wait to be attended). Urgency is defined as that clinical situation with the capacity to generate deterioration or danger to the health or life of the patient, depending on the time elapsed between its appearance and the establishment of an effective treatment, which determines a healthcare episode with significant intervention needs in a short period of time. There are currently six triage systems or models systematically structured into 5 levels.

Although simple in concept, the practice of triage is challenging due to time pressure, the limitations of available information, the various medical conditions of the patients, and a great reliance on intuition on the part of the professionals who perform it. which conditions a great variability in it. On the other hand, almost half of adult ED visits nationwide are classified as level 3 in a 5-level structured triage system, which makes level 3 a heterogeneous group with patients with diverse pathologies, in which triage is not capable of accurately differentiating them, and this inability poses safety risks for the most severely ill patients ("under-triage") and may influence the accuracy and efficiency in resource allocation when patients with low acuity are overrated. Therefore, it seems necessary to develop new triage procedures that allow us to improve their accuracy and reduce inter-individual variability.

TIAGO is a prospective, single-center, observational, comparative study to determine the validity of the Mediktor ® Triage and its effectiveness with respect to the current triage system and the "gold standard" (physician's diagnosis).

DETAILED DESCRIPTION:
Prospective interventional, comparative study to determine the validity of the Mediktor ® Triage and its effectiveness with respect to "Model Andorra of Triage" (MAT) system and the "gold standard" (doctor's diagnosis).

Obtaining informed consent. Participation in the study will be offered to all those patients who attend the Emergency Department of Gynecology and Obstetrics of the Hospital de la Santa Creu i Sant Pau during the study period and who meet the inclusion criteria. An information sheet on the study will also be provided to each patient.

Sequential triage Once the patient's consent has been obtained, the patient will be assessed sequentially in the same triage space. Initially, a nurse from the Gynecology and Obstetrics Service will classify the patient in the triage box using the MAT system according to the usual practice. Then, another professional from the center, trained in the use of the Mediktor Hospital ® tool, and who has not been present in the conventional sorting, will perform the advanced triage in the same space, both professionals being blind to the result of each of the tools. In the event that the first triage performed with MAT gave the investigators an emergency level 1, the triage with the Mediktor tool would not be performed, since in this case the immediate care of the patient would be prioritized.

Attention in the Emergency Service Once the sequential triage is completed, the patient will return to the Gynecology and Obstetrics Emergency Room. The patient's care will be performed according to usual clinical practice, following the triage assessment performed with the MAT system.

Data recovery and entry in Data Recovery Form (DRF) All data of the study variables will be retrieved from the emergency report issued in the area of Gynecology and Obstetrics Emergencies and will be entered in an electronic DRF for further analysis and processing.

Evaluation of Effectiveness

Main evaluation variables Level of triage assigned by MAT, Level of triage assigned by Mediktor Hospital

Secondary evaluation variables

* Affiliation variables (administrative): Date of birth, sex, residence, financing, date and time of arrival in the emergency room or administrative record, form of arrival in the emergency room (own foot, ambulance, etc.…), reason for the urgency ( common illness, traffic accident, school…).
* Triage variables: Triage date and time, triage duration time, coded clinical reason for consultation, readmission within 72 hours, readmission reason, triage level, number of reevaluations, triage level of each reevaluation.
* Care variables: date and time of the emergency room visit, request for additional test, type of additional test, analytical parameters requested (if applicable), diagnosis according to International Classification of Diseases (ICD) (primary and secondary), most important procedures performed, patient admission > 24h), date and time of admission, urgent surgery, time of stay in the emergency room (LOS) which is the time that the patient remains in the emergency room from the time of admission to the hospital until the patient is discharged or hospitalized. Number of patients admitted to the hospital and number of patients discharged. Number of emergency consultations / revisits in the first 72 hours after discharge.
* Variables of discharge: circumstance of discharge or reason for emergency discharge (home discharge, hospital admission, transfer to another center, voluntary discharge, escape, exit…), identification of the transfer center, date and time of discharge, date and time of administrative discharge, departure transport, cause of success, time spent in emergencies, registration canceled

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years
* Understand and accept the study procedures
* Sign the informed consent.

Exclusion Criteria:

* Not being able to understand the nature of the study and/or the procedures to be followed
* Not signing the informed consent
* Be under 18 years of age
* Emergency level 1 through current triage system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with equivalence between emergency triage classifications | 3 days
  Correspondence of emergency grading between Advanced IA Triage Tool (Mediktor Hospital) and the current triage system.

SECONDARY OUTCOMES:
Number of patients with the same diagnosis on advanced triage tool and emergency discharge report (gold-standard) | 3 days
  Assess the correlation between the pre-diagnosis provided by the advanced triage tool and the diagnosis offered by the physician in the emergency discharge report.
Number of patients with good correlation between complimentary tests requested by the advanced triage tool with gold-standard | 3 days
  Assess the correlation between the complementary tests proposed by the advanced triage tool and those requested by the doctors during the emergency room visit, following the care protocols of the center.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Estadella Tarriel, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie results in a publication will be available once the data analysis is completed and the publication have been published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data will be available once the study is published . It will be available for 5 years after publication date.
Access Criteria: Requests will be reviewed by Primary Investigator.

REFERENCES:
- [Background] Mueller B, Kinoshita T, Peebles A, Graber MA, Lee S. Artificial intelligence and machine learning in emergency medicine: a narrative review. Acute Med Surg. 2022 Mar 1;9(1):e740. doi: 10.1002/ams2.740. eCollection 2022 Jan-Dec. PMID 35251669
- [Background] Berlyand Y, Raja AS, Dorner SC, Prabhakar AM, Sonis JD, Gottumukkala RV, Succi MD, Yun BJ. How artificial intelligence could transform emergency department operations. Am J Emerg Med. 2018 Aug;36(8):1515-1517. doi: 10.1016/j.ajem.2018.01.017. Epub 2018 Jan 4. No abstract available. PMID 29321109
- [Background] Raita Y, Goto T, Faridi MK, Brown DFM, Camargo CA Jr, Hasegawa K. Emergency department triage prediction of clinical outcomes using machine learning models. Crit Care. 2019 Feb 22;23(1):64. doi: 10.1186/s13054-019-2351-7. PMID 30795786
- [Background] Levin S, Toerper M, Hamrock E, Hinson JS, Barnes S, Gardner H, Dugas A, Linton B, Kirsch T, Kelen G. Machine-Learning-Based Electronic Triage More Accurately Differentiates Patients With Respect to Clinical Outcomes Compared With the Emergency Severity Index. Ann Emerg Med. 2018 May;71(5):565-574.e2. doi: 10.1016/j.annemergmed.2017.08.005. Epub 2017 Sep 6. PMID 28888332
- [Background] Moreno Barriga E, Pueyo Ferrer I, Sanchez Sanchez M, Martin Baranera M, Masip Utset J. [A new artificial intelligence tool for assessing symptoms in patients seeking emergency department care: the Mediktor application]. Emergencias. 2017 Dic;29(6):391-396. Spanish. PMID 29188913
- [Background] Kuriyama A, Urushidani S, Nakayama T. Five-level emergency triage systems: variation in assessment of validity. Emerg Med J. 2017 Nov;34(11):703-710. doi: 10.1136/emermed-2016-206295. Epub 2017 Jul 27. PMID 28751363
- [Background] Julian-Jimenez A, Palomo de los Reyes MJ, Lain Teres N. [Coment on the original article: modelo predictor de ingreso hospitalario a la llegada al servicio de Urgencias]. An Sist Sanit Navar. 2012 Sep-Dec;35(3):493-6; author reply 497-9. doi: 10.23938/ASSN.0113. No abstract available. Spanish. PMID 23296233
- [Background] Elias P, Damle A, Casale M, Branson K, Churi C, Komatireddy R, Feramisco J. A Web-Based Tool for Patient Triage in Emergency Department Settings: Validation Using the Emergency Severity Index. JMIR Med Inform. 2015 Jun 10;3(2):e23. doi: 10.2196/medinform.3508. PMID 26063343
- [Background] Storm-Versloot MN, Ubbink DT, Kappelhof J, Luitse JS. Comparison of an informally structured triage system, the emergency severity index, and the manchester triage system to distinguish patient priority in the emergency department. Acad Emerg Med. 2011 Aug;18(8):822-9. doi: 10.1111/j.1553-2712.2011.01122.x. PMID 21843217
- [Background] Moll HA. Challenges in the validation of triage systems at emergency departments. J Clin Epidemiol. 2010 Apr;63(4):384-8. doi: 10.1016/j.jclinepi.2009.07.009. Epub 2009 Oct 28. PMID 19875271